CLINICAL TRIAL: NCT05522751
Title: Limbic Pallidum Deep Brain Stimulation for the Treatment of Severe Alcohol Use Disorder
Brief Title: Deep Brain Stimulation for Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khaled Moussawi (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Khaled Moussawi, Assistant Professor of Psychiatry, Neurology, and Bioengineering, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY22030036
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AUD DBS (Experimental): This is a single arm study. Participants will undergo baseline medical and psychiatric assessments, cognitive and behavioral testing, and positron emission tomography (PET) imaging. One to two weeks later, participants will undergo neurosurgical implantation of DBS electrodes in the limbic pallidum and a neurostimulator. Four weeks after DBS system implantation, the DBS system will be turned ON and the stimulation parameters optimized. Participants will be followed biweekly then monthly for repeat comprehensive assessments.
  Interventions: Device: DBS

INTERVENTIONS:
Device: DBS — Bilateral DBS electrodes will be implanted into the limbic pallidum of participants with severe alcohol use disorder and advanced but compensated liver disease.

SUMMARY:
The purpose of this clinical study is to investigate the safety, tolerability, and feasibility of Deep Brain Stimulation (DBS) of the limbic pallidum in participants with severe alcohol use disorder (AUD) who have advanced but compensated liver fibrosis.

DETAILED DESCRIPTION:
Participants with severe AUD will undergo baseline medical and psychiatric assessments, cognitive and behavioral testing, and positron emission tomography (PET) imaging. One to two weeks later, participants will undergo neurosurgical implantation of DBS electrodes in the limbic pallidum and a neurostimulator. Four weeks after DBS system implantation, the DBS system will be turned ON and the stimulation parameters optimized. Participants will be followed biweekly then monthly for repeated comprehensive assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (all genders) 21 to 75 years old.
2. Severe primary Alcohol Use Disorder (AUD) (>= 6 Diagnostic and Statistical Manual-5 AUD criteria) with or without other substance use disorders.
3. Participants are seeking treatment for their AUD (participants receiving medications or other therapy for AUD are eligible).
4. Participants have insight into their alcohol use disorder (score >26 on the recognition subscale of the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES V.8)).
5. Participant has advanced compensated alcohol-associated liver disease (ALD). Compensated is defined as asymptomatic per clinical evaluation (by hepatologist or internist). Advanced is defined as fibrosis stage >= 3; if not previously diagnosed, fibrosis stage >= 3 will be diagnosed with liver elastography using a liver stiffness cutoff >=15kiloPascal
6. AUD is treatment refractory: unable to achieve sustained remission (>12 months) over the past 5 years, despite treatment attempts, with at least one treatment attempt involving completed residential or outpatient treatment program with pharmacotherapy, behavioral therapy, or both.
7. Stated willingness to comply with all study procedures and availability for the duration of the study.
8. Social support system and stable living arrangement to provide assurances that the subject will adhere to study requirements: family or friends who live with or near the subject, and can provide collateral information, monitor the subject's behavior, support, and encourage the subject to participate in follow-up visits and evaluations. This is evaluated by a neuropsychologist.
9. For females of reproductive potential: use of highly effective contraception for at least 4 weeks prior to DBS surgery and agreement to use such a method during study participation, and after study completion if they elect to keep the DBS system implanted and ON.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Non-English speaking.
3. AUD treatment with another investigational drug or other intervention within 3 months.
4. History of primary psychosis or Bipolar I disorder per the psychiatric evaluation or Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders-5 measure.
5. History of severe personality disorder that could interfere with study participation (e.g., antisocial personality disorder) per the psychiatric evaluation, neuropsychological evaluation, or Structured Clinical Interview for the Diagnostic and Statistical Manual-5 measure.
6. Intelligence quotient <75 as measured by Wechesler Abbreviated Scale of Intelligence (evaluated by a neuropsychologist).
7. History of suicidal attempts in the past 5 years or current suicidal thoughts per psychiatric evaluation and Columbia-Suicide Severity Rating Scale (C-SSRS).
8. Decompensated ALD: clinically obvious ascites, hepatic encephalopathy, jaundice episodes, large esophageal varices with or without variceal bleeding, hepatorenal syndrome, per the clinical evaluation (by hepatologist or internist).
9. Coagulopathy: international normalized ratio (INR) > 1.4, activated partial thromboplastin time (aPTT) > 40 s, platelets < 100,000.
10. Current clinically significant medical or neurologic disease that affects brain function (e.g., recent stroke, myocardial infarction, seizures not due to alcohol withdrawal).
11. Clinically significant abnormality on structural brain MRI scan.
12. Life expectancy less than 18 months per the clinical judgement during medical evaluation (e.g., no terminal cancers).
13. Any labeled DBS contraindication or inability to have brain MRI: certain pacemakers, metal in body, inability to undergo awake operation, significant cardiac or other medical risk factors for surgery, infection, and coagulopathy.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Moussawi, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data could be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after study completion.
Access Criteria: all data and information must be de-identified.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 224 potential subjects were prescreened. Most prescreened subjects were not eligible. Around fifteen percent of those who were potentially eligible never followed up or were no longer interested.
Pre-assignment Details: 3 subjects consented and were enrolled. One subject was a screen-fail and was not implanted with the device.
Period: Overall Study
Arm/Group | AUD DBS
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | AUD DBS
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events (Safety and Tolerability)
Description: This will be evaluated based on number and seriousness of adverse events associated with DBS implantation and stimulation (e.g., infection, bleeding, cognitive or behavioral side effects).
Time Frame: 4-52 weeks
Measure: Number; unit: Adverse Events
Arm/Group | AUD DBS
Number analyzed (Participants) | 2
Adverse Events
  Serious Adverse Events | 1
  Other Adverse Events | 1

2. Primary Outcome: Recruitment (Feasibility)
Description: This will be evaluated based on number of participants recruited and enrolled in the study between study start date and primary completion date.
Time Frame: 0-71 weeks
Population: 224 potential participants were pre-screened for recruitment.
Measure: Count of Participants; unit: Participants
Arm/Group | AUD DBS
Number analyzed (Participants) | 224
Participants | 3

3. Primary Outcome: Proportion of Completed Assessments (Feasibility)
Description: This will be evaluated based on the average percentage of evaluations completed across participants during the study duration out of total required assessments to measure the participants' adherence to the study protocol.
Time Frame: 4-52 weeks
Measure: Mean (Full Range); unit: Percent of total assessments
Units Other Than Participants: Evaluations
Arm/Group | AUD DBS
Number analyzed (Participants) | 2
Number analyzed (Evaluations) | 66
Percent of total assessments | 100 [100 to 100]

4. Secondary Outcome: Overall Functioning
Description: Overall function and disability will be measured using standardized questionnaire World Health Organization Disability Assessment 2.0 (WHODAS2.0) score before and after DBS activation (raw score 0-180, higher is worse). The focus of analysis was limited to the 6-month timepoint.
Time Frame: 6 months
Measure: Number; unit: score on a scale
Arm/Group | AUD DBS
Number analyzed (Participants) | 1
score on a scale
  Baseline | 1.61
  6 months | 1.5

5. Secondary Outcome: Alcohol Use - Percent Days Abstinent
Description: assessment of alcohol use will be measured through percent days abstinent (PDA) at baseline (pver preceding 6 months) and at 6 months after DBS activation. PDA at baseline is assessed over the preceding 180 days. PDA at 6 months post-DBS activation is assessed over the preceding 30 days.
Time Frame: 6 months
Measure: Number; unit: percentage of days
Arm/Group | AUD DBS
Number analyzed (Participants) | 1
percentage of days
  Baseline | 14.6
  6 months | 81

6. Secondary Outcome: Alcohol Use - Drinks Per Drinking Day
Description: assessment of alcohol use will be measured through drinks per drinking day (DDD) before and after DBS activation. The focus of analysis was limited to the 6-month timepoint. DDD at baseline is assessed over the preceding 180 days. DDD at 6 months post-DBS activation is assessed over the preceding 30 days.
Time Frame: 6 months
Measure: Number; unit: drinks per drinking day
Arm/Group | AUD DBS
Number analyzed (Participants) | 1
drinks per drinking day
  Baseline | 10.49
  6 months | 5

7. Secondary Outcome: Target Engagement
Description: This will be assessed by measuring the percent change in brain metabolism with 18fluoro-Deoxy-Glucose (FDG) PET scans before and after DBS activation. The timepoint 4 weeks post-surgery was excluded because breath alcohol test was positive on that day.
Time Frame: 6 months
Measure: Number; unit: percentage of cerebellar activity
Arm/Group | AUD DBS
Number analyzed (Participants) | 1
percentage of cerebellar activity
  Limbic pallidum change in activity at 6 months relative to baseline | -7
  Ventral striatum change in activity at 6 months relative to baseline | -13
  OFC change in activity at 6 months relative to baseline | -14

8. Other Pre Specified Outcome: Cue Reactivity Craving Score
Description: To measure subjective craving after presentation of alcohol or neutral pictorial cues pre and post DBS. Craving is reported using a visual analog scale (VAS) between 0 and 100, where 100 indicates very high craving; the cue reactivity craving score is calculated as the difference in craving scores after alcohol vs. neutral pictures.
Time Frame: 6 months
Measure: Number; unit: score on a scale
Arm/Group | AUD DBS
Number analyzed (Participants) | 1
score on a scale
  Baseline | 73.06
  6 months | -3

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | AUD DBS
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUD DBS (N=2)
Intracranial hemorrhage during surgery (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUD DBS (N=2)
surgical wound pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment was halted after the SAE occurrence in one subject. Only one subject completed the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: Study protocol (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT05522751/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT05522751/SAP_001.pdf
  • Informed Consent Form: informed consent form (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05522751/ICF_002.pdf